CLINICAL TRIAL: NCT04214184
Title: Biomarkers and Altered Metabolic Pathways During Sleep Loss
Brief Title: Biomarkers of Increased Free Living Sleep Time
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Christopher Depner, Assistant Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 133959
Record Dates: First submitted 2019-12-17; First posted 2020-01-02 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Sleep Deprivation; Insufficient Sleep Syndrome; Sleep Wake Disorders
MeSH Terms: conditions — Sleep Deprivation; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Participants with habitual insufficient sleep schedules will complete a 4-week increased sleep duration intervention targeting the recommended 7 hours of sleep per night.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Increased Sleep Duration Intervention (Experimental): Following baseline assessments, participants will complete a 4-week increased sleep duration intervention followed by one night of sleep in the lab on this increased sleep duration schedule. In the morning, participants will have blood collected for metabolomics analyses and complete oral glucose tolerance testing
  Interventions: Behavioral: Increased sleep duration

INTERVENTIONS:
Behavioral: Increased sleep duration — Participants will increase their nightly time in bed by 2 hours per night for 4 weeks to target the recommended 7 hours of sleep per night.

SUMMARY:
This protocol will increase sleep duration in participants who maintain less than 6 hours sleep per night, to target the recommended 7 hours of sleep per night. The focus of this study is determine how increasing nightly sleep duration in these individuals who maintain less than 6 hours sleep per night changes their plasma metabolome and insulin sensitivity. The primary outcome will examine changes in branched-chain amino acids and the secondary outcome will examine changes in insulin sensitivity. The investigators will also determine if changes in plasma metabolites can be used as a biomarker to discriminate between adequate versus insufficient sleep.

DETAILED DESCRIPTION:
Impaired sleep affects millions of people each year representing an important public health issue. This project will utilize metabolomics approaches to identify potential mechanisms underlying increased cardiometabolic risk associated with insufficient sleep and to identify potential biomarkers in the blood that respond to insufficient sleep. Investigators will conduct a controlled in-laboratory insufficient protocol where participants will sleep in the lab for one night with sleep timing based on their habitual insufficient sleep schedule. In the morning, plasma will be collected for metabolomics analyses and participants will complete an oral glucose tolerance test for insulin sensitivity analyses. Participants will then complete a 4 -week increased sleep duration intervention targeting the recommended 7 hours of sleep per night. Following this intervention participants will again sleep in the lab for one night on their new sleep schedule. In the morning, plasma will be collected for metabolomics analyses and participants will complete an oral glucose tolerance test for insulin sensitivity analyses. Investigators anticipate these findings will be the first step in developing biomarkers of impaired sleep under free-living sleep conditions, and to determine how such biomarkers relate to insulin sensitivity changes associated with sleep loss.

ELIGIBILITY:
Inclusion Criteria:

1. 18-35 years old; men and women

   a. Equal numbers of women and men will be included.
2. Body Mass Index (BMI) of > 18.5 and <24.9.
3. Inactive to habitual moderate physical activity level (<5 days of exercise per week).
4. Sleep/wake history: habitual sleep duration less than 6 hours per night.
5. Altitude history: Potential participants must have lived at Denver altitude or higher for at least 3 months.

Exclusion Criteria:

1. Any clinically significant unstable medical or surgical condition within the last year (treated or untreated).
2. Any clinically significant psychiatric condition, as defined by DSM-IV-TR. I
3. Any clinically significant sleep disorder.
4. Use of prescription medications/supplements within one month or need of these medications at any time during the study.
5. Symptoms of active illness (e.g., fever).
6. Uncorrected visual impairment
7. History of shift work in prior year or travel more than one time zone in three weeks prior to study.
8. Participants must be entirely drug-free of illicit drugs, medications, nicotine and herbal products for one month prior to study.
9. Blood donation in the 30 days prior to inpatient study.
10. Ovulating women will be selected on the basis of a history of regular menstrual cycle ranging in length from 25-32 days with a maximum of three days variation month-to-month. They will have no history of prior gynecological pathology, be at least 1 year post-partum, not breast-feeding and not pregnant (HCG pregnancy test at screening and upon admission to the inpatient protocol).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolomics-branched chain amino acids change from baseline | Morning fasted blood will be collected for analyses at baseline and after the four week increased sleep duration intervention.
  Investigators will measure the abundance of the branched chain amino acids (valine, leucine, isoleucine) in plasma at baseline and at post intervention.
Insulin Sensitivity change from baseline | Oral glucose tolerance testing will take about 3 hours to complete, and will be tested at baseline and after the four week increased sleep duration intervention.
  Investigators will measure insulin sensitivity using the oral glucose tolerance test in the morning after overnight sleep assessments in the lab, at baseline and after the four week increased sleep duration intervention.

SECONDARY OUTCOMES:
Untargeted Metabolomics change from baseline | Morning fasted blood will be collected for analyses at baseline and after the four week increased sleep duration intervention.
  Investigators can detect relative abundance of ~4,000 plasma metabolites. A combination of metabolites that can discriminate between adequate versus insufficient sleep will be identified as a potential biomarkers of insufficient sleep in free-living adults.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Depner, Principal Investigator — University of Utah
Locations (1):
- Sleep Wake Center--University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data generated from the proposed work that is presented in a peer reviewed journal will be uploaded, de-identified, into the Metabolomics Data Repository and Coordinating Center (DRCC) (U01) through UCSD; http://www.metabolomicsworkbench.org/nihmetabolomics/datasharing.html. In addition, .raw data that is presented in a peer reviewed journal will be archived indefinitely and made available upon request.
Time Frame: Data will become available upon publication in peer-reviewed journals and will be made available indefinitely.
Access Criteria: Active membership and username are required to access the raw metabolomics data on Metabolomics Workbench.